CLINICAL TRIAL: NCT06503471
Title: A Clinical Research on SCLife®-UT hUC-MSCs Advanced Therapy Medicinal Products (hUC-MSCs ATMPs) for Patients With Thin Endometrial Infertility
Brief Title: SCLife®-UT hUC-MSCs Advanced Therapy Medicinal Products (hUC-MSCs ATMPs) for Patients With Thin Endometrial Infertility
Status: Suspended | Phase: Phase 1 | Type: Interventional
Why Stopped: Lack of financial support
Sponsor: Sclnow Biotechnology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SCLnow-NE-01
Record Dates: First submitted 2024-07-02; First posted 2024-07-16 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-12

CONDITIONS: Infertility, Female
MeSH Terms: conditions — Infertility, Female

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: randomize double-blind
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- stem cell and collagen transplantation group (Experimental): Human Umbilical Cord Mesenchymal Stem Cells
  Interventions: Biological: human umbilical cord mesenchymal stem cell complex collagen
- control group (Active Comparator): collagen transplantation
  Interventions: Biological: human umbilical cord mesenchymal stem cell complex collagen; Procedure: intrauterine injection

INTERVENTIONS:
Biological: human umbilical cord mesenchymal stem cell complex collagen — 1 * 10^7 cells (2ml)
Procedure: intrauterine injection — intrauterine injection with human umbilical cord mesenchymal stem cell (19#iSCLife®-UT); total 1 time
  Arms: control group

SUMMARY:
To explore the therapeutic effect and safety of human umbilical cord mesenchymal stem cells on thin endometrial infertility and to explore whether human umbilical cord mesenchymal stem cells using collagen as the carrier can promote endometrial growth, reduce the recurrence rate of intrauterine adhesion, increase the clinical pregnancy rate, improve the pregnancy outcome, and study its safety.

DETAILED DESCRIPTION:
This is a random, open label, and self-control experiment. 24 patients are selected and sign consent forms, then divided into two groups. Doctors collect the basic information of patient (including age, BMI, mental condition, vital sign, history of disease, pharmaco-history, and so on.), evaluate the symptom of thin endometrial infertility (menstrual conditions, uterine cavity form, pregnancies).

All patients receive laboratory and image examination as baseline. Then, cell treatment will be given based on the clinical protocol. Doctors have follow-up visit on 1, 3, 6, 12 month after treatment, and do efficacy evaluation.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged 20 to 39 years with primary or secondary infertility who have received ivf embryo transfer treatment and have been frozen at least 4 good quality embryos (good quality embryos defined as 7-9C / ⅱ 0 or 4BC or more blastocysts and ≥2 grade ⅰ embryos or 4BC or more blastocysts)
2. Once above 2 times under hysteroscopy surgery adhesions, uterine cavity form has returned to normal, with normal menstrual cycle or at least a cycle high-dose estrogen replacement therapy for more than 12 days (> 4 mg/day, maximum dose of more than 8 mg/day), after treatment the biggest endometrial thickness of 7 mm or less or upper middle period of endometrial thickness of 7 mm or less on average; Or received assisted reproductive therapy, after at least 4mg/ day of estrogen, colony stimulating factor, aspirin, sildenafil and other drugs, unknown maximum endometrial thickness ≤7mm or average endometrial thickness ≤7mm in middle and upper segment; The maximum endometrial thickness in luteal phase was less than 6mm
3. 18kg/m2< body mass index (BMI) <24 kg/m2
4. Voluntarily participate and sign the informed consent
5. Negative coV-19 nucleic acid test

Exclusion Criteria:

1. Uncured sexually transmitted diseases
2. Participate in other clinical investigators within 3 months
3. Serum pregnancy tested positive
4. Coagulopathy or other diseases of the blood system
5. Severe heart disease, unstable angina attack, cardiac insufficiency of grade III or above, acute myocardial infarction and/or old myocardial infarction, hypertension was diagnosed according to the guidelines for prevention and treatment of hypertension in China (2010 edition)
6. Patients with active genital tuberculosis
7. Patients with immune system disorders
8. Diseases related to pregnancy outcome (any) : Untreated hydrosalpinx, untreated uterine polyp, untreated uterine infection, phase III ~ Ⅳ endometriosis and adenomyosis of the uterus, ovarian cyst > 4 cm, uterine fibroids > 2 cm in diameter, multiple muscle intramural myoma, and submucosal fibroids, cesarean section incision site benign tumor prognosis, basin celiac > 4 cm, pituitary tumors and malignant tissues and organs tumors
9. Abnormal uterine bleeding
10. Severe liver and kidney function injury, namely, blood alanine aminotransferase (ALT) and aspartate aminotransferase (AST) were 2.5 times higher than the upper limit of normal value, and blood creatinine (Cr) and urea nitrogen (BUN) were 2 times higher than the upper limit of normal value
11. The researcher considers that she is not suitable for this study

Ages: 20 Years to 39 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 24 (Estimated)
Dates: Start 2025-12-31 (Estimated); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Pregnancy outcome | 12 months
  Pregnancy status is tracked for pregnancy rate, clinical pregnancy rate, ongoing pregnancy rate, miscarriage rate and live birth rate.

CONTACTS AND LOCATIONS:
Locations (1):
- Changsha Reproductive Medicine Hospital (Changsha Ning 'er Maternity Hospital), Changsha, Hunan, China

IPD SHARING:
Plan to Share IPD: No